CLINICAL TRIAL: NCT00596258
Title: A Two-Stage Phase 2 Study Of Dose-Intense 4,4'-Dihydroxybenzophenone-2,4-Dinitrophenyl-Hydrazone (A-007) Topical Gel in the Treatment of High-Grade Squamous Intraepithelial Lesions (HSIL) of the Cervix
Brief Title: A Two-Stage Phase 2 Study Of A-007 Topical Gel in High-Grade Squamous Intraepithelial Lesions (HSIL)
Acronym: TG-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tigris Pharmaceuticals (Industry)
Responsible Party: Anne White, Tigris Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-003
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Cervical Intraepithelial Neoplasia; Uterine Cervical Dysplasia
Keywords: Cervical Intraepithelial Neoplasia (CIN); High-grade Cervical Intraepithelial Neoplasia; High-grade Squamous Intraepithelial Lesions (HSIL); Human Papilloma Virus (HPV); High-Grade Cervical Intraepithelial Lesions (CIN 2/3)
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — 4,4'-dihydroxybenzophenone-2,4-dinitrophenylhydrazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A-007 (Experimental): Single arm open label
  Interventions: Drug: A-007

INTERVENTIONS:
Drug: A-007 — applied topically for two 28-day cycles of 14 consecutive days of treatment each to the uterine cervix

SUMMARY:
A-007 is an investigational therapy which may be effective in the treatment of pre-cancerous cervical dysplasia (abnormal cell growth). The purpose of this study is to evaluate the safety and efficacy of A-007, when used to treat high-grade cervical dysplasia.

DETAILED DESCRIPTION:
This is a non-randomized, two-stage phase II study with pathological response rate as the primary objective. Following biopsy confirmation of CIN 2/3 within the last 12 weeks, women will treat themselves with gel applied to the cervix via an intravaginal applicator. Patients will apply gel once daily for 14 consecutive days of a 28-day cycle for 2 cycles.

Women will return to clinic for safety assessments, colposcopy, cytology, and virologic and immunologic testing (see schedule of events in attachment TG-003.01 for visit intervals).

Following the two cycles of treatment with A-007, treating physicians will perform a LEEP at the month 4 visit. The investigator is responsible for ensuring that the LEEP is conducted according to the procedures and guidelines of their institution.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* The patient or her authorized representative must sign and date an Ethical Review Board-approved informed consent document. All aspects of the protocol must be explained and written informed consent obtained.
* Patients must have histologic proof of CIN 2/3 disease documented within the last 12 weeks. If patient is enrolled using prior local biopsy, local slides and pathology report must be sent to the central laboratory. Patient may be enrolled into the study based on local laboratory results of CIN 2/3 and will not be discontinued if central laboratory results differ.
* Cervical swabs must test positive for high risk HPV (by Hybrid Capture 2). If the patient tests negative for high risk HPV and has proof of CIN 2/3, the patient should be retested one additional time for high-risk HPV.
* Patients must have a Hgb ≥ 9 g/dl, a peripheral WBC ≥ 3000 mm3 and platelet counts ≥100,000 mm3.
* Normal hepatic and renal functions - AST and ALT <2.5 x ULN and creatinine <1.5 x ULN, respectively.
* Females of childbearing potential must use one of the following birth control methods during the study (until performance of the LEEP at month 4): oral, implantable, injectable contraceptives; abstinence (celibacy). Contraceptive sponges, IUD, vaginal contraceptive rings, spermacides, sponges, condoms, or partner's vasectomy are not acceptable methods of birth control.

Exclusion Criteria:

* Patients with CIN 1 or with invasive squamous cell carcinoma (SCC).
* CIN appearing to involve the endocervix, as assessed colposcopically
* CIN not amenable to adequate colposcopic follow-up evaluations, i.e. unsatisfactory colposcopy.
* CIN 3 involving more than two cervical quadrants on colposcopy.
* Patients treated for cervical SIL within the past year.
* Patients who have had a LEEP performed in the past 12 months
* Patients with other malignancy (except non-melanoma skin) within the past 5 years.
* Patients with any chronic, active infections (including HIV) other than HPV.
* Patients with known clinically relevant immunological deficiency.
* Concurrent treatment with cytotoxic, radiation, or immuno-stimulative therapy, or with systemic corticosteroids at a dose >5 mg/d of prednisone (or its equivalent).
* Participation in another investigational medication trial concurrently or within 30 days, or prior administration of a prophylactic HPV vaccine or participation in an HPV vaccine trial. Treatment within the last 30 days with a medication that has not received regulatory approval at the time of study entry.
* Concomitant use of topical vaginal medications.
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.
* History of allergy or hypersensitivity to cosmetics, toiletries, or other topical or dermatologic products.
* Pregnant or lactating females who are nursing and will not consent to cease nursing.
* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Patients with known menstrual irregularity that is not resolved with cycling on hormonal contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Determine overall pathological response (complete and partial, based on independent review at month 4) of A-007 when applied topically for two 28-day cycles of 14 consec. days of treatment each to the uterine cervix of women with HSIL [CIN 2/3]. | Over the course of the trial

SECONDARY OUTCOMES:
Determine the local tolerability and systemic safety of A-007. | over the course of the trial
Evaluate the effects of A-007 gel treatment on human papillomavirus (HPV) eradication. | over the course of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Aqua, MD, Principal Investigator — Visions Clinical Research; Mark H Einstein, MD, Principal Investigator — Montefiore Medical Center-Weiler Division; Cynthia J Goldberg, MD, Principal Investigator — Visions Clinical Research-Tucson; Robert Pfeffer, MD, Principal Investigator — Robin Black OGNP, Costa Mesa California; Stephanie Blank, MD, Principal Investigator — NYU School of Medicine
Locations (5):
- United States (5):
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Robin Black OGNP, Costa Mesa, California
  - Visions Clinical Research, Boynton Beach, Florida
  - NYU School of Medicine, New York, New York
  - Montefiore Medical Center-Weiler Division Dept of OB/GYN & Women's Health, The Bronx, New York

REFERENCES:
- [Background] Morgan LR, Thangaraj K, LeBlanc B, Rodgers A, Wolford LT, Hooper CL, Fan D, Jursic BS. Design, synthesis, and anticancer properties of 4,4'-dihydroxybenzophenone-2,4-dinitrophenylhydrazone and analogues. J Med Chem. 2003 Oct 9;46(21):4552-63. doi: 10.1021/jm0301080. PMID 14521417
- [Background] Morgan, LR, Hooper, CL, Rodgers, AH, LoRusso, P, Eilender, DE and Culotta, VA. 4,4'-Dihydroxybenzophenone-2,4-dinitrophenyl-hydrazone (A-007): A CD4+ T-Lymphocyte Modulator Useful in the Treatment of Advanced Cancer. Chemotherapy - accepted 2005.
- [Background] Morgan, LR, Hooper, CL, Rodgers, AH Culotta, V et al. 4,4'-Dihydroxy benzophenone -2,4-dinitrophenylhydrazone (A-007) A Modulator of CD45+ T Lymphocytes in HPV Infected Anogenital Epithelium. In: HPV Vaccines and Immune Therapy, Cambridge, United Kingdom, 2003